CLINICAL TRIAL: NCT02383108
Title: A Two-arm, Phase 2/3 Multicentre, Open-label, Randomised Study Evaluating Safety and Antiviral Effect of Current Standard Antiretroviral Therapy Compared to Once Daily Integrase Inhibitor Administered With Darunavir/Ritonavir (DRV/r) in HIV-1 Infected, Virologically Suppressed Paediatric Participants.
Brief Title: Strategy for Maintenance of HIV Suppression With Once Daily Integrate Inhibitor+Darunavir/Ritonavir in Children
Acronym: SMILE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); MRC CTU at UCL (Unknown); PHPT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMILE (PENTA 17); ANRS1 52 (Other: France Agency for research on AIDS and viral hepatitis)
Record Dates: First submitted 2015-02-19; First posted 2015-03-09 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care group (SOC) (Active Comparator): triple anti-retroviral therapy including 2 NRTIs + boosted PI/NNRTI
  Interventions: Drug: SOC
- DTG+DRV/r (Experimental): NRTI-sparing regimen: Once daily integrase inhibitor (INSTI) + darunavir/ritonavir (DRV/r)
  Interventions: Drug: DTG +DRV/r

INTERVENTIONS:
Drug: DTG +DRV/r — NRTI-sparing regimen: Once daily integrase inhibitor (INSTI) + darunavir/ritonavir (DRV/r)
  Arms: DTG+DRV/r
Drug: SOC — Standard of care (continuing triple anti-retroviral therapy including 2 NRTIs + boosted PI/NNRTI)
  Arms: Standard of Care group (SOC)

SUMMARY:
A two-arm, Phase 2/3 multicentre, open-label, randomised study evaluating safety and antiviral effect of current standard antiretroviral therapy compared to once daily integrase inhibitor administered with darunavir/ritonavir (DRV/r) in HIV-1 infected, virologically suppressed paediatric participants.

DETAILED DESCRIPTION:
A two arm parallel group, non-inferiority, open-label, multi-centre, randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected children aged ≥ 12 years old and weighing ≥40kg* at the screening visit
2. Aged 12 to < 18 years old**
3. Parents or guardians, and children where appropriate, willing and able to give informed consent and to adhere to the protocol
4. Children must have all HIV-1 RNA viral loads <50c/mL for at least 12 months with a minimum of two separate results before screening.
5. Children on a 3-drug PI/r or NNRTI containing regimen for at least 24 weeks
6. Children/parents/guardians prepared to switch if randomised to once daily integrase inhibitor + DRV/RTV arm
7. Children and parents prepared to restart the current ART regimen after simplification if viral load restart criteria are met (see Section 5.5)
8. Be affiliated or beneficiary to Health Social security scheme (in countries where this is mandatory)

   * Initially enrolment will be of participants ≥ 12 years old and ≥40kg only. DTG 50 mg will be supplied by ViiV Healthcare.

     * As more data become available on younger children, a protocol amendment is planned to include younger children and/or lower weight bands.

Exclusion Criteria:

1. Receiving or requiring agents with interactions with DRV, RTV, or any once daily integrase inhibitor (Appendix 14)
2. Evidence of resistance to DRV or integrase inhibitors (for participants in clinical sites where resistance testing is standard of care)
3. Previous exposure to integrase inhibitors for more than 2 weeks
4. Intercurrent illness (randomisation can take place after the illness resolves)
5. Creatinine ≥ 1.8ULN or ALT ≥ 5ULN or ALT ≥ 3ULN and bilirubin ≥2ULN at screening.
6. Patients with severe hepatic impairment or unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
7. Diagnosis of tuberculosis and on anti-tuberculosis treatment (children can be enrolled after successful tuberculosis treatment)
8. Hepatitis B or Hepatitis C co-infection
9. Pregnancy or risk of pregnancy in girls of child-bearing potential unless committed to taking effective contraception
10. History or presence of known allergy or some other contraindication to the study drugs or their components as described in the SmPC

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2016-06; Primary Completion 2020-08 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with HIV-1 RNA ever ≥ 50 c/mL (confirmed within 4 weeks) | at any time up to week 48

SECONDARY OUTCOMES:
Percentage of patients with HIV-1 RNA < 50 c/mL | at week 48
Percentage of patients with HIV-1 RNA ≥ 50 c/mL | at week 24
Percentage of patients withHIV-1 RNA ≥ 400c/mL | at week 24 and week 48
Percentage of patients with any grade 3 or 4 clinical adverse events (particularly lipodystrophy); any grade 3 or 4 laboratory adverse events | over 48 weeks
All grade 3 or 4 laboratory adverse events | over 48 weeks
Any adverse event at least possibly related to study drugs or leading to treatment modifications | over 48 weeks
Occurrence of new resistance mutations | over 48 weeks
Changes in CD4 (absolute and percentage) | from baseline to weeks 24 and 48
Change in ART (defined as any change from the ART regimen at randomisation) | at week 0
New or recurrent CDC/WHO stage C or severe stage B event or death | over 48 weeks
Blood lipids | over 48 weeks
Adherence as measured by questionnaire and visual analogue scale | over 48 weeks
Acceptability and quality of life over 48 weeks as assessed by patient completed questionnaires | over 48 weeks
Tanner scales (in participants aged over 8 years) | over 48 weeks
Date of first menses | over 48 weeks
Height | Over 48 weeks
Weight | over 48 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- Hospital Garrahan, Buenos Aires, Argentina
- France (2):
  - Centre Hospitalier Andrée Rosemon, Cannes
  - CHU Hôtel Dieu - Nantes, Nantes
- Hospital General Mexico, Mexico City, Mexico
- Portugal (2):
  - Hospital de Dona Estefânia - CHLC, Lisbon
  - Centro Materno-Infantil de Norte, Porto
- South Africa (2):
  - FAM-CRU, Cape Town
  - PHRU, Soweto
- Spain (6):
  - Hospital San Joan de Deu, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Getafe, Madrid
- Switzerland (3):
  - Inselpital Bern, Bern
  - Kantonsspital St Gallen, Sankt Gallen
  - Kinderspital Zurich, Zurich
- Thailand (6):
  - Prapokklao Hospital, Chanthaburi
  - Nakornping Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Kalasin hospital, Kalasin
  - Khonkaen hospital, Khon Kaen
  - Phayao hospital, Phayao
- Uganda (2):
  - Baylor, Kampala
  - JCRC, Mbarara
- Ukraine (2):
  - Kiev, Kiev
  - Kryvyi Rih, Kryvyi Rih
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Hospital, Bristol
  - Evelina Children Hospital, St Thomas's Hospital, London
  - King's College Hospital, London

REFERENCES:
- [Derived] Compagnucci A, Chan MK, Saidi Y, Cressey TR, Bamford A, Riault Y, Coelho A, Nolan A, Chalermpantmetagul S, Morkunaite G, Amuge P, Musiime V, Violari A, Cotton M, Kekitiinwa AR, Kaudha E, Groenewald M, Liberty AA, Kanjanavanit S, Volokha A, Bologna R, Pavia Ruz N, Prieto Tato L, Paioni P, Marques L, Reliquet V, Niehues T, Welch SB, Ford D, Giaquinto C, Gibb DM, Babiker A, Ramos Amador JT; SMILE-PENTA17-ANRS 152 Trial Group. Nucleoside/nucleotide reverse transcriptase inhibitor sparing regimen with once daily integrase inhibitor plus boosted darunavir is non-inferior to standard of care in virologically-suppressed children and adolescents living with HIV - Week 48 results of the randomised SMILE Penta-17-ANRS 152 clinical trial. EClinicalMedicine. 2023 Jun 2;60:102025. doi: 10.1016/j.eclinm.2023.102025. eCollection 2023 Jun. PMID 37304494